CLINICAL TRIAL: NCT05725226
Title: Comparison Between Standard Vs Small Sized Double J Stent On Urological Symptoms Following RIRS And URSL: A Prospective Randomized Controlled Trial
Brief Title: Comparison Between 6Fr Vs 4Fr Double J Stent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tribhuvan University, Nepal (Other)
Responsible Party: Principal Investigator, Prajwal Khatiwada, Resident Doctor in General Surgery Department, Tribhuvan University, Nepal
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PKhatiwada
Record Dates: First submitted 2023-01-13; First posted 2023-02-13 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Renal Stone; Ureter Stone
MeSH Terms: conditions — Nephrolithiasis; Ureterolithiasis

STUDY DESIGN:
Intervention Model Description: Participants are assigned to study where two groups of treatments, Group 1 (6 Fr) and Group 2 (4Fr), are given so that Group 1 will receive 6Fr Double J stent after endourological stone fragmentation and Group 2 will receive 4Fr Double J stent after endourological stone fragmentation.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 : 6Fr (Active Comparator): Procedure: RIRs/URSL Confirmation of Renal/ Ureteric Stone with CT Urography Preanesthetic Check up and SterileUrine Culture obtained prior to surgery Perioperative Care: Inj. Ceftriaxone 1gm IV stat dose , RIRS/ URSL performed using LASER Holmium lithotripsy 6Fr Double J stent is inserted to maintain the ureteric patency USSQ score obtained on Post operative Day 3, Day 7 and on the day of stone removal (Day 14) USG Abdomen and Pelvis is done on post operative Day 30 to confirm stone clearance.
  Interventions: Device: Double J Stent 6Fr x 26cms
- Group 2: 4Fr (Experimental): Procedure: RIRs/URSL Confirmation of Renal/ Ureteric Stone with CT Urography Preanesthetic Check up and SterileUrine Culture obtained prior to surgery Perioperative Care: Inj. Ceftriaxone 1gm IV stat dose , RIRS/ URSL performed using LASER Holmium lithotripsy 4Fr Double J stent is inserted to maintain the ureteric patency USSQ score obtained on Post operative Day 3, Day 7 and on the day of stone removal (Day 14) USG Abdomen and Pelvis is done on post operative Day 30 to confirm stone clearance.
  Interventions: Device: Double J Stent 4Fr x26cms

INTERVENTIONS:
Device: Double J Stent 6Fr x 26cms — Surgery will be performed by expert Urologist.
  Arms: Group 1 : 6Fr
Device: Double J Stent 4Fr x26cms — Surgery will be performed by expert Urologist.
  Arms: Group 2: 4Fr

SUMMARY:
Double J (DJ) Stenting is a commonly done procedure in endourology to ensure ureteric patency following Urological Interventions. DJ stents are available in various sizes. This study is focused on comparing two different sizes of DJ Stents, one standard sized 6Fr and other small sized 4Fr. DJ stents are uncomfortable to the patients and few studies have indicated that small size of stents are might be less troublesome. Through this study we plan to establish a relation between different symptoms and size of DJ stents. Study will be conducted at Tribhuvan University Teaching Hospital (TUTH),Maharajgunj.All adults with sterile urine culture prior to stenting will be taken into consideration. Informed consent will be taken and two randomized groups of 6Fr and 4Fr will be formed and data entry done in MS Excel and analysis done by SPSS. The study is expected to take duration of 12months. Ureteral Stent Symptom Questionnaire (USSQ) will evaluate the symptoms on third day and seventh day of stent placement and on Day of stent removal. We expect 4Fr stent to be superior to 6Fr for reduction of stent related symptoms.

DETAILED DESCRIPTION:
The concept of the endoscopic access to the renal collecting systems for the diagnosis and treatment of upper urinary tract diseases was firstly introduced by V. Marshall who first described in 1964 the navigation in the renal pelvis with a rudimental flexible fiberscope. Retrograde intrarenal surgery (RIRS) by means of flexible ureterorenoscopes (fURSs) is considered one of the first-line treatment options for the active removal of renal stones. Ureteroscopic Lithotripsy (URSL) with the holmium laser is an effective and safe method for treating ureterolithiasis. After RIRS, one of the technical aspect is the placement of a double-J stent. The underlying rationale of ureteric stent is to allow the urinary flow to bypass internal or external obstructions, which impair its drainage. 'Double-J' refers to the most common type of stent design that was initially introduced by Finney in 1978. The term 'double-J' refers to the 'J' shape of each end of the stent, which is designed to anchor the stent and prevent its displacement. The mean size of normal ureter is 1.8mm with a standard deviation of 0.9 mm. The standard size for double J stents is typically 6 Fr. Few studies have been done comparing standard 6Fr and smaller sized DJ stent. One study published in March 2018 has shown 4Fr stent superior to 5Fr and 6Fr stent. A Randomised Control Trial (RCT) published in July 2018 has shown 4.8 Fr stent superior to 6Fr stent. To assess ureteral stent-related symptoms, Joshi et al. described and validated the Ureteral Stent Related Symptom Questionnaire (USSQ) in 2003. This self-administered questionnaire includes questions in six sections: urinary symptoms, body pain, general health, work performance, sexual matters, and additional problems. The total score is the sum of all questions. This questionnaire can define and compare stent-related symptoms.

DJ stent cause significant side effects. Dysuria, urinary frequency and urgency were reported by 40%, 50% and 55% of the patients, respectively. Flank pain, gross hematuria and fever was reported by 32%, 42% and 15% respectively. Anxiety and sleep disturbance were reported by 24% and 20% respectively, and 45% of patients reported impairment in their quality of life. Decreased libido was reported by 45%, and sexual dysfunction by 42% of men and 86% of women. With few studies showing small sized DJ stent causing less symptoms that standard 6Fr stents; our study aims to ascertain whether the previous studies were in line to change the standard size of DJ stent from 6Fr to smaller size, possibly 4Fr. 6Fr DJ stent is commonly used in our center. This study is aimed to compare standard size of DJ stent with small size in TUTH.

All cases of urinary tract stones requiring endourologic intervention will be sampled for study and cases meeting the inclusion criteria will be randomized via simple random sampling and computer generated numbers enclosed in a sealed envelope opened just prior to surgery, into two groups: Group A 6Fr and Group B 4Fr. All cases will receive a single dose of ceftriaxone intraoperatively. RIRS will be done using Ureteral Access Sheath (UAS) 9.5-11.5 Fr. DJ Stent 4Fr or 6Fr will be used and length of DJ Stent will be 26cm. Stent will be removed on the 14th postoperative day. Symptoms will be assessed on day 3, day 7 and on the day of stent removal. Stone Clearance will be assured after 1 month with ultrasonography of abdomen.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18yrs
* Informed Consent
* Sterile Urine culture prior to surgery

Exclusion Criteria:

* Bilateral DJ stenting
* Pregnancy
* Ureteral Strictures
* Complicated Surgery: Trauma, Bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2023-04-07 (Actual); Primary Completion 2023-12-21 (Actual); Study Completion 2023-12-21 (Actual)

PRIMARY OUTCOMES:
To compare Ureteral Stent Symptom Questionnaire (USSQ) scores following 6Fr vs 4Fr Double J stenting | 14 days
  Ureteral Stent Symptom Questionnaire score will be obtained by requesting the participants to fill the questionnaire. The questionnaire will be filled on post operative Day 3, Day 7 and Day 14. The maximum possible score is 169 and minimum score is 33. Higher score indicates poor performance of Double J stent.

SECONDARY OUTCOMES:
To analyze the demographic pattern of patients undergoing URSL and RIRS in TUTH | 1day, on the date of admission
  All demographic data are entered prior to surgery.
To compare the pain score, urinary symptoms, general health, sexual symptoms and work performance following 6Fr and 4Fr Double J Stenting | 14 days
  Ureteral Stent Symptom Questionnaire score is the sum of the scores of pain symptoms, urinary symptoms, general health symptoms, work performance symptoms and sexual symptoms. All these components will also be analyzed separately.
To compare stone clearance following 6Fr and 4Fr Double J stenting | Post operative day 30
  Stone Clearance will be confirmed by ultrasonography done post operatively on Day 30.

CONTACTS AND LOCATIONS:
Overall Officials: Pawan Rj Chalise, MCh Urology, Study Chair — Head of Department, Department of Urology and Kidney Transplant Surgery, TUTH
Locations (1):
- Tribhuvan University Teaching Hospital (TUTH), Institute of Medicine, Kathmandu, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: No